CLINICAL TRIAL: NCT05746234
Title: A Pilot Feasibility Study for an Emotion Regulation Skills Training (ER4ALL) for Students in Higher Education
Brief Title: Emotion Regulation For All (ER4ALL) Study
Acronym: MASHUP1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cyprus (Other)
Collaborators: VU University of Amsterdam (Other); University of Crete (Other); Eotvos Lorand University (Other)
Responsible Party: Principal Investigator, Prof. Georgia Panayiotou, Dr. Georgia Panayiotou, Professor of Clinical Psychology, Department of Psychology and Center for Applied Neuroscience, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MashUP_FeasibilityRCT1
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Emotion Regulation
Keywords: Emotion regulation, Mental Health, Socio-Emotional Learning
MeSH Terms: conditions — Emotional Regulation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will use a pre-post design with a multi-case study approach to evaluate the feasibility and implementation of the ER intervention in four university settings.
  A mixed-methods design will be used to determine the feasibility and acceptability of the "ER4ALL" course.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music-Based ER module (Experimental): The program will involve the following modules: a) VALUES & SETTING GOALS FOR ENHANCING MOTIVATION, b) MODULE 2. UNDERSTANDING EMOTIONS, c) MODULE 3. MINDFUL EMOTION AWARENESS AND RELAXATION, d) MODULE 4. THINKING FLEXIBLY, e) MODULE 5. COUNTERING INAPPROPRIATE BEHAVIORS.
  The rationale of the training was built based on the framework of Unified Protocol (Barlow, et al. 2018) and training activities were selected and adapted from a compilation of foundational works on contemporary evidence-based approaches, (i.e. Cognitive Behavioral approach, Acceptance and Commitment approach, and Dialectical Behavior approach). Activities were adapted using core components of music-based interventions (Dingle & Fay, 2016; McFerran, 2016; Saarikallio, 2019) with emphasis on emotion recognition in music, regulation of stress and negative emotions through active music listening, and self-reflective awareness of emotional responses to music.
  Interventions: Behavioral: Emotion Regulation Course
- Standard ER module (Active Comparator): Participants will receive the same training modules in the same chronological order as the music-based group. The only difference is that modules will be mainly text/language based (instead of using music methodologies).
  Interventions: Behavioral: Emotion Regulation Course

INTERVENTIONS:
Behavioral: Emotion Regulation Course — Each module contains a) the session outline, b) review of previous session's homework, c) theoretical background and module's rationale, d) skills activities, and e) homework assignment.
  Each group will attend five 1.5-hour sessions with their allocated instructor. Participants in both groups will receive the same training modules in the same chronological order. For consistency across modalities, participants will receive an instructor's manual containing the core material for facilitating the ER4ALL training, and a companion students' workbook with supporting information and activities.
  Other Names: ER4ALL course

SUMMARY:
In the present study, the investigators aim to examine the feasibility of a classroom-based emotion regulation skills training within a tertiary curriculum.

The primary objective of this study is to assess the acceptability and feasibility of the "ER4ALL", a brief course for enhancing emotion regulation skills for students in higher education.

The secondary objective of this study is to collect preliminary evidence for beneficial effects in increasing students' acquired knowledge on adaptive emotion regulation, thus improvement on general psychological wellbeing.

A two-arm pilot RCT will be conducted in University of Cyprus.

DETAILED DESCRIPTION:
Entering Higher Education (HE) marks a turning point for youth learning to function as independent adults, something that can be both exciting and challenging. Students are confronted with a considerable number of changes to manage (e.g. high academic expectations, making new relationships, making independent decisions), for which they may be psychosocially unfamiliar or uncomfortable.

Several studies have indeed shown that rising levels of difficulty in socio-emotional adaptation for students in HE, is linked to decreased levels of engagement and completion rates. On the other hand, the acquisition of psycho-social skills, seems to have a positive effect on students' academic achievement, resilience, employability and thriving in life.

A current challenge for HE Institutions is to ensure that during their studies, their future graduates, will have the opportunity to develop psycho-social skills, for effective management of challenges, which extend beyond academic contexts and outcomes throughout the life span in domains such as success in work, positive interpersonal relationships, and better mental health and overall well-being.

Further examination of the potential impact of integrating empirically supported transversal components that derive from empirical research (e.g. emotion regulation skills), is needed. In addition to that, since the focus is on a university-wide student population, it would be useful to further investigate whether the standard mode of delivery (in which learning capacity, language ability, and executive functions are considered essential ingredients for program success), fits well to student population with diverse learning styles, academic performance or learning abilities, such as language skills (listening, reading, speaking and writing), executive skills (e.g. sustain attention) or cognitive processes such as memory and abstract thinking. A growing literature pinpoints to the potential of incorporating art-based methodologies, such as music which is characterized by personalized methods and has shown promising effects on its effectiveness for inclusive educational practices. Music is a promising means that can afford opportunities for learning not afforded by other modalities. Collectively, music holds the potential to address life-long needs for young adults, by infusing culturally appropriate practices that can be easily integrated into the young adults' everyday experiences at the level of their abilities. Music interventions have been linked to improvements in mental and physical capacities in various settings and populations. Research findings additionally support that music can be used as a tool for emotion regulation by reducing stress and stimulate cognitive processes such as attention, learning and memory. Taking into account the above, it is of great interest to develop and investigate how different modalities, such as music-based methodologies, can alter the effectiveness of existing empirically supported approaches, such as emotion regulation skills training.

The primary objective of this study is to gain insight into the acceptability and feasibility of the "ER4ALL", a brief course for enhancing emotion regulation skills for students in higher education. The secondary objective of this study is to collect preliminary evidence for beneficial effects in increasing students' acquired knowledge on adaptive emotion regulation, thus improvement on general psychological functioning.

The specific objectives of the study are to:

1. Determine feasibility and acceptability of the "ER4ALL" course.

   1. To estimate feasible recruitment and refusal rates.
   2. To measure key outcome domains such as completion rates, missing data, students-reported measures of social satisfaction (both qualitative and quantitative).
   3. To determine the acceptability of course resources and factors influencing this (e.g. diverse learning styles or abilities).
2. Compare the effectiveness between two "ER4ALL" modalities: standard language-based mode Vs. music-based mode.

   1. To explore preliminary differences on acceptability.
   2. To explore preliminary differences on associated changes in acquired knowledge and psychological functioning.

ELIGIBILITY:
Inclusion Criteria - People who are enrolled as students in the university

Exclusion criteria

- No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the course | up to 10 weeks
  At post-training, principal researchers involved in the development and delivery of the intervention in each site, will complete Structured Assessment of FEasibility (SAFE; Bird et al. 2014), a standardised measure of the feasibility of complex interventions (Bird et al. 2014). The SAFE measure comprises 16 items grouped into two sub-scales: Blocks (8 items) and Enablers (8 items). SAFE guidelines recommend that reviewers attend to the individual items of the scale, instead of using summary scores, since items have unequal weight. Τhe tool has shown excellent interrater reliability (k = 0.84, 95% CI 0.79-0.89) and test-retest reliability (k = 0.89, 95% CI 0.85-0.93).
Acceptability of the course | up to 10 weeks
  At post-training, all participants will complete a course satisfaction/acceptability questionnaire. The questionnaire will consist of two parts: In part A (quantitative) students will be asked several Likert-scale questions, while part B (qualitative) while contain open-ended response questions relating to their experience, satisfaction, and the challenges/enablers associated with design and implementation of the course. Qualitative data from open-ended questions will be considered alongside the quantitative measures to assess the feasibility of the intervention. The feasibility and acceptability of the intervention will be evaluated, using multiple primary endpoints such as:
  1. Adherence (Total registrations, Attendance Rates, Homework Adherence, Dropouts)
  2. Course acceptability and satisfaction ratings
  3. Training preference.

SECONDARY OUTCOMES:
Emotion Beliefs Questionnaire | up to 10 weeks
  The EBQ (Becerra, Preece, & Gross, 2020) is a 16-item self-report measure of beliefs about emotions. Based on Ford and Gross's (2019) theoretical framework, the EBQ assesses two main categories of beliefs about emotions: beliefs about the controllability of emotions and beliefs about the usefulness of emotions. These beliefs are assessed for negative emotions and positive emotions. Four subscale scores and three composite scores are designed to be derived from the measure, with higher scores indicating more maladaptive beliefs about emotions (i.e., stronger beliefs that emotions are uncontrollable and useless). The scale has demonstrated good concurrent validity (EBQ scores correlated significantly in expected ways with various scores from other measures of beliefs about emotions), as well as validity and internal consistency in its initial validation (α = .88; Becerra, Preece, & Gross, 2020).
Acceptance and Action Questionnaire-II | up to 10 weeks
  Acceptance and Action Questionnaire-II (AAQ-II; Bond et al., 2011) is a 7-item measure of psychological flexibility rated on a 7-point scale (Cronbach's α = 0.84). It assesses the ability to be fully present in the moment and adjusting behaviors based on the situational demands, personal values and goals. Higher total score means less flexibility.
Psyflex | up to 10 weeks
  Psyflex (Gloster, et al 2021) is a 6-item self-report questionnaire designed to measure in a brief and context-sensitive manner all six facets of psychological flexibility based on Acceptance and Commitment Theory. Items are rated on a scale from 5 ("very often") to 1 ("very rarely") and then summed. Higher scores represent higher psychological flexibility. Confirmatory Factor Analysis confirmed a one-factor structure with excellent reliability (Raykov's r = 0.91).
Positive Mental Health Scale (PMH-scale) | up to 10 weeks
  The 9-item PMH-scale was developed in order to provide a brief, uni-dimensional and person-centered instrument to assess positive mental health (Lukat et al. 2016). The PMH-scale assesses mainly emotional, but also psychological and social aspects of well-being. Participants respond to statements such as "I am in good physical and emotional condition" or "I manage well to fulfill my needs" on a scale ranging from 0 (I disagree) to 3 (I agree). Higher scores reflect greater positive mental health. Psychometric testing confirmed the scale to be a unidimensional self-report instrument with high internal consistency (Cronbach's alpha .82-93), good retest-reliability (r between samples >.74), and good convergent and discriminant validity (e.g. positive correlation with satisfaction with life, r = .75), (Lukat et al. 2016).
Depression Anxiety Stress Scales (DASS-21) | up to 10 weeks
  DASS-21 (Henry, & Crawford, 2005) is a general mental health tool consisting of three scales (7 items per scale) measuring states of depression, anxiety and stress on a 4 point Likert scale (0 'almost always' to 4 'never'). Ηigher scores indicating a greater number of symptoms. The DASS-21 subscales show good internal consistency (Cronbach's α = 0.81- 0.88).
Brief Multidimensional Students' Life Satisfaction Scale-College (BMSLSS-C) | up to 10 weeks
  BMSLSS-C (Zullig et al. 2009) is a brief version of MSLSS addressing circumscribed aspects of college students´ life. In specific it consists of 9 items, one for each of the following life satisfaction domains LSS (family, friends, school, self, and living environment, romantic relationships, physical appearance, and work). Higher scores represent higher college satisfaction. The scale has shown an acceptable reliability (a=.80), and criterion-related validity (significantly correlated with the CDC HRQOL-14 and Social Isolation Scale in predicted directions) in its initial validation.
University Student Learning Disabilities Questionnaire | up to 10 weeks
  University Student Learning Disabilities Questionnaire (Glenn et al., 1997) is a screening evaluation of behavioral and cognitive characteristics exhibited by college students in learning and testing situations. A higher score represents higher Learning Difficulties. During its initial validation, a logistic regression analysis verified the predictive capability of the final subset of items, which has also shown high test-retest reliability (.83; Glenn et al., 1997).

OTHER OUTCOMES:
Participants characteristics | up to 10 weeks
  Questions concerning sociodemographic characteristics (age, gender, education level, academic field, preference for randomization condition, previous history / previous use of mental health services).
Fidelity | up to 10 weeks
  To support the establishment of competency, instructors will be invited to:
  1. Fill procedural fidelity checklists after each session, to self-assess whether or not the training objectives were met as outlined in training and in the guidebook. Fidelity total scores will be reviewed.
  2. An external evaluator will attend 2 randomly selected sessions and rate the sessions using fidelity checklists.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided